CLINICAL TRIAL: NCT02262910
Title: A Phase 1 Study of ES414 in Patients Wtih Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study of ES414 in Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aptevo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 401
Record Dates: First submitted 2014-09-26; First posted 2014-10-13 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: metastatic castration-resistant prostate cancer; CRPC
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ES414 (Experimental): Cohorts 1-3 of the dose escalation stage of the study (Stage 1) will test weekly doses of 0.2 mcg/kg to 2 mcg/kg. Cohorts 4-9 of the dose escalation stage of the study (Stage 1) will test continuous infusion at flat doses of 25 mcg to 300 mcg per day delivered continuously over 24 hours. The maximum tolerated dose from Stage 1 of the study will be further examined in Stage 2. Patients in cohorts 1-3 will receive ES414 weekly via intravenous (IV) infusion during the first three 28-day cycles and then on Day 1 and 15 of each subsequent cycle until disease progression, intolerable toxicity occurs, or the patient withdraws consent. Patients in cohorts 4-9 will receive ES414 as a continuous IV infusion for 6 months until disease progression, intolerable toxicity occurs, or the patient withdraws consent.
  Interventions: Biological: ES414

INTERVENTIONS:
Biological: ES414 — ES414 is a novel humanized bispecific antibody which is designed to treat mCRPC by redirecting T-cell cytotoxicity against prostate cancer cells expressing prostate-specific membrane antigen (PSMA).

SUMMARY:
The study will be conducted in 2 Stages. The primary objective of Stage 1 of the study is to identify the maximum tolerated dose (MTD) of ES414 administered intravenously to patients with mCRPC. Secondary objectives are to evaluate the tolerability, pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity, cytokine response, and clinical activity of ES414.

The primary objective of Stage 2 of the study is to evaluate the clinical activity of ES414 in patients that have or have not received prior chemotherapy. Secondary objectives are to further characterize the safety profile, PK, PD, and immunogenicity of ES414.

DETAILED DESCRIPTION:
Stage 1 - Dose Escalation: The dose escalation stage of the study will test weekly doses of 0.2 mcg/kg to 300 mcg/kg over 9 dose levels (cohorts). Cohorts 1 to 3 consist of single patients and Cohorts 4 - 9 will consist of a minimum of 3 patients; an additional 3 patients may be added to the cohort if adverse events possibly related to ES414 or dose-limiting toxicities (DLT) occur. The next dose cohort will only enroll after the patient(s) in the current dose cohort have completed the first cycle of dosing (4 weeks) with no significant adverse events or DLTs. Six patients will be enrolled at the maximum tolerated dose (MTD) and this dose will be used for Stage 2.

Stage 2 - Expansion: The continuous intravenous infusion MTD dose regimen will be further examined in 2 expansion cohorts; the first cohort are patients that have received prior chemotherapy, such as docetaxel for mCRPC, and the second cohort are those that have not received prior chemotherapy for mCRPC. Serum samples will be collected for serial PK assessment for ES414 drug levels and antibody formation. Response will be assessed every 2 months during the first 6 months of treatment and then every 3 months until progression of mCRPC, intolerable side effects, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate. No evidence of neuroendocrine differentiation or small cell features.
* Surgically or medically castrated, with testosterone ≤ 50 ng/dL (≤ 1.7 nmol/L).
* Progressive prostate cancer by either serum PSA levels, soft tissue or bone disease as defined by the PCWG2 criteria.
* In Stage 1, patients may or may not have received prior chemotherapy for mCRPC. In Stage 2, patients will be enrolled into two cohorts based on whether or not they have received prior chemotherapy for mCRPC. Any prior chemotherapy must have been completed ≥ 4 weeks prior to administration of ES414. Additionally, in countries where abiraterone or enzalutamide are commercially available, patients in Stage 1 and 2 must have progressed on abiraterone and/or enzalutamide prior to study entry.
* ECOG ≤ 1
* Life expectancy > 6 months per investigator
* Adequate hematologic, renal, and hepatic parameters

Exclusion Criteria:

* Any chemotherapy, sipuleucel-T, or investigational drug in prior 4 weeks, or abiraterone or enzalutamide in prior 2 week
* Any radiation therapy in prior 2 weeks
* Any prior therapy targeted against PSMA
* History of seizures
* History of central nervous system metastasis
* History of nephrotic syndrome
* Spot urine total protein:creatinine ratio >1,000 mg/gm
* Planned palliative procedures for alleviation of bone pain
* Active infection requiring treatment with systemic anti-infectives or major surgery in prior 4 weeks.
* Any prednisone (or equivalent corticosteroids) use within 2 weeks of study entry
* Chronic immunosuppressive therapy
* Known history of HIV, hepatitis B, or hepatitis C infection
* Evidence of severe or uncontrolled systemic diseases
* History of bleeding disorders or thromboembolic events in prior 3 months

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of ES414 | during first 28 days of treatment
  Identify the maximum tolerated dose in dose-escalation stage (Stage 1) by assessment of dose-limiting toxicities

SECONDARY OUTCOMES:
Safety Profile of ES414 | Patients will be followed for the duration of treatment, an expected average of 6 months, and for 28 days following last treatment
  The safety profile of ES414 will be assessed by monitoring incidence and severity of adverse events
Maximum Serum Drug Concentration (Cmax) | Pre- and post-infusion at least weekly during first 28-day cycle, and on Days 1 and 15 of subsequent cycles for an expected duration of 6 months, and for up to 8 weeks following last treatment
  Blood samples will be obtained from all patients for determination of the maximum serum concentration of ES414.
Area under the concentration versus time curve (AUC) | Pre- and post-infusion at least weekly during first 28-day cycle, and on Days 1 and 15 of subsequent cycles for an expected duration of 6 months, and for up to 8 weeks following last treatment
  Blood samples will be obtained from all patients for determination of the AUC of ES414.
Elimination half-life (T1/2) | Pre- and post-infusion at least weekly during first 28-day cycle, and on Days 1 and 15 of subsequent cycles for an expected duration of 6 months, and for up to 8 weeks following last treatment
  Blood samples will be obtained from all patients for determination of the T1/2 of ES414.
Immune-Related Response Criteria (irRC) | Baseline and 6 months
  Investigator measurements of target lesions
Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Baseline and 6 months
  Investigator measurements of target lesions
Pharmacodynamics of ES414 | Patients will be followed for the duration of treatment, an expected average of 6 months, and for 28 days following last treatment
  Blood samples will be collected from all patients and evaluated by flow cytometry for changes in lymphocytes
PSA Response | Baseline and 6 months
  Blood samples will be collected from all patients and tested for PSA
Circulating Tumor Cells | Patients will be followed for the duration of treatment, an expected average of 6 months, and for 28 days following last treatment
  Blood samples will be collected from all patients and evaluated for the number of circulating tumor cells
Immunogenicity of ES414 | Patients will be followed for the duration of treatment, an expected average of 6 months, and for 8 weeks following last treatment
  Blood samples will be collected from all patients and tested for antibody formation to ES414.

CONTACTS AND LOCATIONS:
Overall Officials: Scott C Stromatt, MD, Study Director — Aptevo Therapeutics
Locations (7):
- United States (4):
  - University of California, San Francisco, California
  - Roswell Park Cancer Institute, Buffalo, New York
  - Central Texas Veterans Health Care System, Temple, Texas
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington
- Australia (3):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria